CLINICAL TRIAL: NCT01209975
Title: Retinal Vascular Reactivity in Response to Isoxic Hypercapnia in Subjects With Newly Diagnosed Glaucoma
Brief Title: Retinal Vascular Reactivity in Subjects With Newly Diagnosed Glaucoma Before and After Selective Laser Trabeculoplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Dr. Chris Hudson, Department of Ophthalmology and Vision Science
Other Study IDs: SLT-blood flow study
Record Dates: First submitted 2010-06-29; First posted 2010-09-28 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Glaucoma
Keywords: blood flow; glaucoma; SLT
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- untreated glaucoma patients: We will evaluate the blood flow before and after Selective Laser Trabeculoplasty in patients with primary open angel glaucoma.
  Interventions: Procedure: Selective Laser Trabeculoplasty

INTERVENTIONS:
Procedure: Selective Laser Trabeculoplasty — Patient will have selective laser trabeculoplasty as the first treatment for glaucoma. This treatment will be dictated clinically, since we do not assign the interventions.

SUMMARY:
The purpose of this study is to assess retinal blood flow and vascular reactivity in patients with newly diagnosed primary open angle glaucoma pre- and post-primary Selective Laser Trabeculoplasty(SLT). Canon Laser Blood Flowmeter will be used for the assessment of retinal blood flow.

DETAILED DESCRIPTION:
We previously found that vascular reactivity improved after short term treatment with dorzolamide drops. It is not clear whether this improvement was a direct effect of the medication or secondary effect of the decrease in IOP. We would like to see the change of vascular reactivity before and after SLT, which will decrease the intraocular pressure without pharmacologic effect.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-75 years (Male or Female)
2. Best corrected visual acuity of at least 20/40
3. No previous treatment for glaucoma
4. Ametropia less than ±6.0 DS and ±2.5 DC)
5. Non-smoker
6. No cardiovascular/respiratory disorders

Exclusion Criteria:

1. Past history of diabetes and cerebrovascular accident
2. Vascular occlusive disease affecting the ocular circulation such as: diabetic retinopathy, retinal vein occlusion and retinal artery occlusion
3. Previous intraocular surgery
4. Ocular media opacities limiting the use of the imaging tests

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with untreated primary open angle glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
blood flow | before and two-week after SLT
  The Canon Laser Blood Flowmetry will be used to assess the retinal blood flow.

SECONDARY OUTCOMES:
Intraocuclar pressure | before and two-week after SLT
  Intraocular pressure (IOP) will be measured by Goldmann applanation tonometry.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Hudson, PhD, Principal Investigator — University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Venkataraman ST, Hudson C, Rachmiel R, Buys YM, Markowitz SN, Fisher JA, Trope GE, Flanagan JG. Retinal arteriolar vascular reactivity in untreated and progressive primary open-angle glaucoma. Invest Ophthalmol Vis Sci. 2010 Apr;51(4):2043-50. doi: 10.1167/iovs.09-3630. Epub 2009 Nov 11. PMID 19907031